CLINICAL TRIAL: NCT04276818
Title: Use of Platelet-Rich Plasma in Second-Degree Superficial Burns; Multicentric Prospective Randomized Study
Brief Title: Use of Platelet-rich Plasma in Second-degree Superficial Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, Principal Investigator, Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBU Konya EAH
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Burns Degree Second
Keywords: PRP; Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Active Comparator): Second-degree superficial burn group treated with PRP
  Interventions: Procedure: PRP group
- conventional treatment group (Active Comparator): second-degree superficial burn group treated with cream containing silver sulfadiazine
  Interventions: Procedure: conventional treatment group

INTERVENTIONS:
Procedure: PRP group — Demonstrating the effectiveness of dressing with PRP in the treatment of second-degree burns
  Arms: PRP group
Procedure: conventional treatment group — The effectiveness of conventional dressing containing silver sulfadiazine in the treatment of burns will be compared with the method of dressing with PRP.
  Arms: conventional treatment group

SUMMARY:
Platelet-rich plasma (PRP) obtained from the patient's blood has been used in many clinical and experimental studies, primarily wound healing, and successful results have been achieved.

PRP has been used in various studies in the treatment of burn wounds, and positive results have been obtained. However, investigators did not find any study or publication about the use of PRP in second-degree superficial burns in our screening.

Investigators planned a prospective randomized controlled and multicenter study to investigate the positive effects of PRP in the treatment of second-degree superficial burn.

DETAILED DESCRIPTION:
The study was planned to be performed between 01.03.2020 and 01.04.2020 in Health Sciences University Konya Training and Research Hospital Burn Unit and Health Sciences University Mogadishu-Somalia Recep Tayyip Erdogan Training and Research Hospital General Surgery Clinics.

Patients hospitalized with a second degree superficial burn and treated with PRP will be included in the study.

Primary purpose: To investigate the effectiveness of platelet-rich plasma in burn treatment Secondary purpose: None. Platelet-rich plasma has recently been used in medicine for the treatment of various diseases.

In our study, patients hospitalized in our clinic with the diagnosis of second-degree superficial burn were randomized and divided into two equal groups. It was planned to treat the first group with PRP, and the second group to be treated with a conventional method of dressing containing silver sulfadiazine cream.

Patients will be given clear and understandable information about the study. Patients who agree to participate in the study will receive a consent form explaining that they have participated in the study voluntarily.

The secretary will do randomization with the help of a computer program. A note stating which group the patient is in will be placed in a closed envelope. A randomization envelope will be opened in each patient before starting treatment.

The primary endpoint of the study was determined as the day when the burn was epithelialized 100%.

Secondary endpoints are the deepening of the wound and the application of other treatment modalities, including surgery, or an infection in the burn area.

In our power analysis, investigators found the number of patients as 80% power and 28 patients with an alpha value of 0.05. Assuming that 10% of patients will be excluded during the study, investigators calculated that a total of 31 patients should be studied.

ELIGIBILITY:
Inclusion Criteria:

* having a second-degree superficial burn
* To be over the age of 16.

Exclusion Criteria:

* Patients under 16
* Patients with a burn of more than 30% of the total body surface area.
* Patients with additional trauma with a burn wound.
* Diabetes mellitus, renal failure requiring dialysis and having decompensated heart disease
* Being pregnant and breastfeeding.
* The patient does not want to participate in the study.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
PRP use in second degree burn treatment | 01.03.2020-30.04.2020
  In the study, the effectiveness of burn treatment in both groups will be determined by recording the day of epithelialization.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not plan to share if it is not necessary

REFERENCES:
- [Background] Venter NG, Marques RG, Santos JS, Monte-Alto-Costa A. Use of platelet-rich plasma in deep second- and third-degree burns. Burns. 2016 Jun;42(4):807-14. doi: 10.1016/j.burns.2016.01.002. Epub 2016 Jan 25. PMID 26822695
- [Background] Grippaudo FR, Carini L, Baldini R. Procutase versus 1% silver sulphadiazine in the treatment of minor burns. Burns. 2010 Sep;36(6):871-5. doi: 10.1016/j.burns.2009.10.021. Epub 2010 Jan 15. PMID 20079572
- [Background] Zheng W, Zhao DL, Zhao YQ, Li ZY. Effectiveness of platelet rich plasma in burn wound healing: a systematic review and meta-analysis. J Dermatolog Treat. 2022 Feb;33(1):131-137. doi: 10.1080/09546634.2020.1729949. Epub 2020 Feb 21. PMID 32048887